

# NON-INTERVENTIONAL (NI) STUDY PROTOCOL

# **Study information**

| Title Protocol number Protocol version identifier Date | Retrospective, non-interventional study to evaluate Chronic Myeloid Leukemia treatment landscape and real-life treatment outcomes in Hungary: analysis of National Health Insurance Fund database B1871064 1.0 16 Nov 2020 |
|---|---|
| Active substance | bosutinib (L01XE14). |
| Medicinal product | bosutinib (Bosulif) |
| Research question and objectives | The <b>objectives</b> of this study are to describe patient demographics, clinical and disease characteristics and treatment patterns of CML in Hungary. The primary endpoint of this study is the overall survival of CML patients treated with tyrosine kinase inhibitors in Hungary. The OS of all enrolled patients, OS by sequence pattern and by the number of treatment lines will be analyzed. |
| | Secondary objectives are description of the treatment length in 1st and later lines, incidence and prevalence of CML, the patient demographics (as age, gender, comorbidities), average number of patients' comorbidities, most frequent comorbidities and patient number with comorbidities at baseline and at different treatment lines by investigated TKI, distribution of the investigated TKI therapies by treatment lines |

| | and the real-life treatment sequences in Hungary. | |
|--------|---------------------------------------------------|--------|
| Author | PPD | MD PPD |
| | PPD | |
| | Hungary | |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 3 |
|---|---|
| 2. LIST OF ABBREVIATIONS | 5 |
| 3. RESPONSIBLE PARTIES | 7 |
| 4. AMENDMENTS AND UPDATES | 10 |
| 5. MILESTONES | 11 |
| 6. RATIONALE AND BACKGROUND | 12 |
| 7. RESEARCH QUESTION AND OBJECTIVES | 13 |
| 3. RESEARCH METHODS | 14 |
| 8.1. Study design | 14 |
| 8.2. Setting | 14 |
| 8.2.1. Inclusion criteria | 15 |
| 8.2.2. Exclusion criteria | 15 |
| 8.3. Variables | 15 |
| 8.4. Data sources | 17 |
| 8.5. Study size | 17 |
| 8.6. Data analysis | 18 |
| 8.7. Limitations of the research methods | 21 |
| 8.8. Other aspects | 22 |
| 9. PROTECTION OF HUMAN SUBJECTS | 22 |
| 9.1. Patient information | 22 |
| 9.2. Patient consent | 22 |
| 9.3. Institutional review board (IRB)/Independent ethics committee (IEC) | 22 |
| 9.4. Ethical conduct of the study | 22 |
| 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 23 |
| 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| 12. REFERENCES | 23 |
| 13. LIST OF TABLES | 24 |
| ANNEX 1 LIST OF STAND ALONE DOCUMENTS | 24 |

| Bosutinib |
|--------------------------------------------|
| B1871064 NON-INTERVENTIONAL STUDY PROTOCOL |
| v1.0 16.11.2020 |

| Λ. | MMEV | 2 | A D | DIT | ION | TAT | ГΤ | NIE | $\cap$ I | 7 ( | 1 / | ľΓ | TI | N | 2 | ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Α | NNEA | | Aυ | וולו | IOT | N A | | INF | υi | < IV | /I /- | ١ | ш | יוע | <br> | _4 |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| 1L | First line treatment |
| 2L | Second line treatment |
| 3L | Third Line |
| AE | Adverse Event |
| BCL-ABL1 | Breakpoint Cluster Region—Abelson fusion gene |
| CCR | Complete Clinical Response |
| CML | Chronic Myeloid Leukemia |
| DSU | Drug Safety Unit |
| ELN | European LeukemiaNet |
| EMA | European Medicine Agency |
| ICD -10 | International Classification of Diseases – 10 <sup>th</sup> revision |
| ICHI | International Classification of Health Interventions |
| IEC | Independent ethics committee |
| IRB | Institutional review board |
| MR | Molecular response |
| NHIF | National Health Insurance Fund |
| NPP | Named Patient Program |
| OS | Overall Survival |
| Ph | Philadelphia |

| TKI | Tyrosine Kinase Inhibitor |
|----------|---------------------------------------------------------|
| TTT code | The code used by NHIF to identify the medicinal product |

# 3. RESPONSIBLE PARTIES

# Principal Investigator(s) of the Protocol

| Name, degree(s) | Job Title | Affiliation | Address |
|---------------------------|-----------|-------------|----------------|
| Prof. PPD<br>MD, PhD, DSc | PPD | PPD | PPD |
| PPD MD, | PPD | PPD | PPD Hugnary |
| PPD<br>MD, PhD | PPD | PPD | PPD<br>Hungary |
| PPD<br>MD | PPD | PPD . | PPD Hungary |
| PPD<br>MD | PPD | PPD | PPD |

#### 4. ABSTRACT

**Study Title**: Retrospective, non-interventional study to evaluate Chronic Myeloid Leukemia treatment landscape and real-life treatment outcomes in Hungary: analysis of National Health Insurance Fund database

**Protocol Version and Date**: Version 1.0; 16 Nov 2020

Primary Author: PPD MD, PPD

Hungary

Rationale and background: Patients, with the diagnosis of chronic myeloid leukemia (CML) nowadays expect a life expectancy close to the average life expectancy, due to the availability of the targeted Bcr-Abl tyrosine kinase inhibitor (TKI) treatments. However, the majority of patients should receive continuous treatment for an indefinite period, even for the rest of their lives. Five TKIs (imatinib, nilotinib, dasatinib, bosutinib, and ponatinib) are available in Hungary in everyday clinical practice.

By the decision of the CML, treatment physicians should take into account the patient's risk classification, comorbidities and patient preferences not only by determining first-line treatment but at therapy switch. Despite the excellent results, half of the patients will eventually fail (due to intolerance or resistance) to first-line treatment, and many may require a second, third, or even additional line of therapy.

Few publications exist on real-world treatment pattern from Western Europe, but there is no such data from Hungary so far. Given the population, genetic, cultural, health condition and health care system differences on country and geographic region level, it is important to investigate real world data regionally.

**Research question and objectives:** The objectives of this study are to describe patient demographics, clinical and disease characteristics and treatment patterns of CML in Hungary.

The **primary endpoint** of this study is the overall survival of CML patients treated with tyrosine kinase inhibitors in Hungary. The OS of all enrolled patients, OS by sequence pattern and by the number of treatment lines will be analysed and displayed on Kaplan-Meier curve.

**Secondary objectives** are description of the treatment length in 1<sup>st</sup> and later lines, incidence and prevalence of CML, the patient demographics (age, gender, comorbidities), average number of patients' comorbidities, most frequent comorbidities and patient number with comorbidities at baseline and at different treatment lines by investigated TKI, distribution of the investigated TKI therapies by treatment lines and the real-life treatment sequences in Hungary.

**Study design:** Retrospective, non-interventional study to evaluate Chronic Myeloid Leukemia treatment landscape and real-life treatment outcomes in Hungary using the database of the National Health Insurance Fund of Hungary

**Population:** All patients treated with TKI based on CML diagnosis between 01 January 2011-30 June 2020.

**Variables:** The variables assessed in this study are patient demographics, clinical characteristics, comorbid conditions, chronic myeloid leukemia treatment history and TKI treatment pattern.

**Data sources:** Prescription claims data, outpatient and inpatient data from the database of the National Health Insurance Fund of Hungary. Hungary provides universal healthcare for its citizens, thanks to the single-payer public system, the NHIF database contains all prescription claims data of all reimbursed medicinal products, all outpatient and inpatient data from all Hungarian patients.

**Study size:** Approximately 1000-1200 patients' data will be analysed.

**Data analysis:** The mathematical algorithm required for analysis is designed and provided by RxTarget Statistical Programming and Analysis Ltd. using SQL programming language based on a preliminary study plan. The algorithm is run by experts at NHIF using primary social security number-level data from selected patients. Anonymized data is provided by NHIF in an aggregated form without any individual identification parameter based on a specific permit, with the strict consideration of data protection rules. Descriptive statistics will be applied for the variables, and no hypothesis is tested.

#### **Milestones:**

| Milestone | Planned date |
|----------------------------|--------------|
| Start of data analysis | Q4 2020 |
| End of data analysis | Q4 2020 |
| First report | Q4 2020 |
| Final study report | Q1 2021 |
| Manuscript for publication | Q3 2021 |

# 5. AMENDMENTS AND UPDATES

None.

# 6. MILESTONES

| Milestone | Planned date |
|----------------------------|--------------|
| Start of data Analysis | Q4 2020 |
| End of data Analysis | Q4 2020 |
| First report | Q4 2020 |
| Final study report | Q1 2021 |
| Manuscript for publication | Q3 2021 |

#### 7. RATIONALE AND BACKGROUND

CML is a neoplastic disease whose genetic and cytogenetic changes play important roles in prognosis and treatment strategies. Philadelphia (Ph) translocation t(9;22)(q34;q11) results the BCL-ABL1 fusion gene causing a constitutively activated tyrosine kinase. The presence of the Philadelphia (Ph) chromosome or the BCL-ABL1 fusion gene is part of the diagnosis of the disease. The course of the disease consists of 3 stages, the chronic, the blast phase and the accelerated phase. In the chronic phase, up to 30-40% of patients are asymptomatic and approximately 85% of patients are diagnosed in this phase. The chronic phase is played to the played phase and the accelerated phase. The chronic phase is part of the diagnosis of the disease consists of 3 stages, the chronic, the blast phase and the accelerated phase. In the chronic phase, up to 30-40% of patients are asymptomatic and approximately 85% of patients are diagnosed in this phase.

According to the international literature the incidence of chronic myeloid leukemia (CML) is 1-1.5 / 100,000 inhabitants per year. Prevalence trend to be 4 times higher than the incidence. The increase in prevalence began with the introduction of tyrosine kinase inhibitors (TKI). Based on the literature data, the average age of patients at diagnosis is 60-65 years, and CML is exceptionally rare in childhood. Slightly more men are affected by this disease than women (1.2-1.3: 1).

The primary goal of the treatment is to achieve complete cytogenetic remission and a significant molecular response. Treatment should be started immediately after diagnosis and the majority of patients should receive continuous treatment for an indefinite period, or even for the rest of their lives to control the malignant disease. TKI treatment should be withheld during pregnancy. Treatment discontinuation may be considered in patients with durable deep molecular response with the goal of achieving treatment free remission.<sup>2</sup>

The prognosis of chronic myeloid leukemia (CML) has changed since the introduction of imatinib in the early 2000's. Survival in CML patients changed and improved drastically with the introduction of imatinib. At the time of diagnosis, patients can expect a normal life expectancy nowdays. With imatinib treatment, 8-10 years survival rates are above 80%, and the cause of death in CML patients is typically unrelated to CML, in most cases related to comorbidities. 4,5

The most effective treatment options are the drugs belonging to the group of tyrosine kinase inhibitors (TKIs), however, allogeneic haematopoietic stem cell transplantation is still the therapeutic option available. First-, second- and third generation tyrosine kinase inhibitors are currently available. The ELN (European LeukemiaNet) 2020 guideline provides guidance for physicians to develop an appropriate treatment strategy.<sup>2</sup>

According to the latest guidelines (ELN 2020), beside the efficacy of the TKIs, the contraindications and typical adverse event profile, early and late toxicity profile of the available TKIs, the risk classification, patient preferences and even the existing comorbidities should be taken into account by designing the treatment plan. The results of the available first- and second-generation TKIs suggest that a more rapid and deeper molecular response can be achieved with second-generation TKIs, however, there is no significant difference in long-term survival between first-generation imatinib and second-generation TKIs (dasatinib, nilotinib, bosutinib).<sup>2</sup>

Close monitoring of the therapeutic response is required and made by regular monitoring BCL-ABL1 levels at specified intervals. Switching the therapy may occur in the case of relapse, resistance to the TKI or intolerable toxicity. As nowadays 5 TKIs are available, patients may receive several lines of TKI therapies. Approximately half of the patients will start 2<sup>nd</sup> line treatment after first line imatinib within 5 years of therapy.<sup>5</sup>

In Hungary bosutinib is accessible for patients within its EMA label since 2013 via individual reimbursement, and via regular reimbursement since 2017 in 2<sup>nd</sup> and later lines. Imatinib the first TKI for CML has been used since 2001, and generics became marketed in 2017. Nilotinib and dasatinib are reimbursed both in first- and second line of CML therapy since 2014-2015.

TKIs are the standard of care in the treatment of chronic phase. Imatinib, nilotinib and dasatinib are currently reimbursed in Hungary as first line treatment. If resistance or intolerance is developed, beside previously listed second generation TKIs even bosutinib or ponatinib are recommended by the national Finance Protocol.<sup>3, 8</sup> Bosutinib is not reimbursed in first line. Ponatinib is available in Named Patient Program (NPP) in later lines.

Few publications exist on real-world treatment pattern from Western Europe<sup>6,7</sup>, but there is no such data from Hungary so far. Given the population, genetic, cultural, health condition and health care system differences on country and geographic region level, it is important to investigate real world data regionally.

## 8. RESEARCH QUESTION AND OBJECTIVES

The objectives of this study are to describe patient demographics, clinical and disease characteristics and treatment patterns of CML in Hungary and evaluate how these key features have changed in investigated time period.

The **primary endpoint is** overall survival of CML patients treated with tyrosine kinase inhibitors in Hungary.

- OS of all enrolled patients
- OS by sequence pattern (where patients meet the inclusion criteria and the available data allows the analysis). Sequence patterns according the actual marketing authorisation of the investigated products are listed in the Table 1.
- OS by the number of treatment lines

## Secondary objectives are

• the incidence and prevalence of CML in Hungary total, and per year during the investigated period

- patient demographics (age, gender) of all enrolled CML patients
- patient comorbidities based on Charlson comorbidity index
  - average number of patients' comorbidities at baseline (start of the 1L treatment) and at different treatment lines (at the point of treatment switch regardless of the TKIs)
  - o most frequent comorbidities for each investigated TKI total and by treatment lines (investigated comorbidities listed in Table 2.)
  - o average number of patients' comorbidities at the start of different treatment lines (1L, 2L, 3L etc) by investigated TKIs regardless of the previous treatment
  - o patient number with 0, 1, 2 or more than 2 comorbidities at the start of different treatment lines (1L, 2L, 3L etc) by investigated TKIs regardless of the previous treatment
- distribution of the investigated TKI therapies by treatment lines: 1L, 2L, 3L, 4L etc.
- description of real-life treatment sequences as listed in the Table 1.
- description of the length of each therapeutic line by investigated TKIs during real-life use and dose-intensity in each treatment line by TKIs

The use of tyrosine kinase inhibitors in the study is on label in accordance with the EMA and the Hungarian marketing authorisation.

## 9. RESEARCH METHODS

## 9.1. Study design

The study is a retrospective, non-interventional study to evaluate Chronic Myeloid Leukemia treatment landscape and real-life treatment outcomes in Hungary using the database of the National Health Insurance Fund of Hungary. The NHIF database is a nationwide insurance system covering close to 100% of the Hungarian population, which collects patient ID and ICD-10 code information about all in- and out-patient visits, as well as about all prescription of drugs which are reimbursed in Hungary. All data are anonymized at data extraction, and we use non-identifiable data at further analyses.

#### 9.2. Setting

In our study, we retrospectively examine the characteristics of CML treatment, treatment patterns, and duration of treatments, focusing on tyrosine kinase inhibitor treatments by analysis on a NHIF database. From 01 January 2011, all patients treated with tyrosine kinase inhibitors (imatinib, dasatinib, nilotinib, bosutinib, ponatinib) will be included in the study

until the date of data closure (expected until 30 June 2020), this is approximately 1000-1200 patients from all Hungarian Hematology centers. Data collection starts 2 years before (01 January 2009). The analysis period, the years of 2009-2010, will be used as reference years in order to detect only the real starting therapies from 2011(Figure 1).

Figure 1. Study design



#### 9.2.1. Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Female and male patients diagnosed with chronic myeloid leukemia
- 2. Patients receiving tyrosine kinase inhibitor therapy under the terms of the current marketing authorization

## 9.2.2. Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Patients receiving TKI for non-CML diagnoses

## 9.3. Variables

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Age | Demographic characteristics | Medical record | Date of birth |
| Sex | Demographic characteristics | Medical record | Male /Female |

| Incidence | Disease<br>characteristic | Medical record | Number of patients<br>newly diagnosed<br>with CML during<br>the defined period |
|---|---|---|---|
| Length of treatment by lines and total | Disease<br>characteristic | Medical record | Time from 1st CML<br>TKI prescription to<br>time to prescription<br>of another CML TKI |
| Prevalence | Disease<br>characteristic | Medical record | Number of all CML patients during the defined study period |
| Overall survival | Disease<br>characteristics | Medical record | Time from first diagnosis of CML until death |
| Comorbidities at baseline | Patient<br>characteristics | Medical record | Comorbidities coded based on the ICD-10 (listed in Table 2.) at the start of first TKI treatment for CML. |
| Comorbidities at different treatment lines | Patient<br>characteristics | Medical record | Comorbidities coded<br>based on the ICD-10<br>(listed in Table 2.) at<br>switch of TKI<br>treatment for CML |
| 2 <sup>nd</sup> line therapy | Treatment characteristic | Medical record | Use of another CML<br>TKI therapy after 1 <sup>st</sup><br>line |
| 1 <sup>st</sup> line therapy | Treatment characteristic | Medical record | 1 <sup>st</sup> prescription of<br>any CML TKI after<br>first CML diagnosis |
| Length of treatment by lines | Treatment characteristics | Medical record | Lengths of treatment analysed in each line |
| Number of treatment lines | Treatment pattern | Medical record | Number of therapy<br>lines used TKI for<br>CML |

| TKI distribution by therapeutic lines | Treatment pattern | Medical record | Distribution of TKI<br>therapies among all<br>patients in the same<br>line of therapy |
|---|---|---|---|
|---|---|---|---|

#### 9.4. Data sources

National Health Insurance Fund's prescribing and in/outpatient database will be used for the analysis. The database is nationwide, electronic and includes all treated patients. From 01 January 2011, all patients treated with tyrosine kinase inhibitors (imatinib, dasatinib, nilotinib, bosutinib, ponatinib) will be included in the study until the date of data closure (expected until 30 June 2020). Data collection starts 2 years before the analysis period, the years of 2009-2010 will be used as reference years in order to detect only the real starting therapies from 2011.

# 9.5. Study size

Approximately 1000-1200 patients' data will be analysed who were treated with TKI (imatinib, dasatinib, nilotinib, bosutinib, ponatinib) for CML between 01 January 2011 until the date of data closure (expected until 30 June 2020) will be included in the study. Data collection starts 2 years before the analysis period, the years of 2009-2010 will be used as reference years in order to detect only the real starting therapies from 2011.

# 9.6. Data management

The mathematical algorithm required for analysis is designed and provided by RxTarget Statistical Programming and Analysis Ltd. using SQL programming language based on a preliminary study plan. The algorithm is run by experts at NHIF using primary social security number-level data from selected patients. Anonymized data is provided by NHIF in an aggregated form without any individual identification parameter based on a specific permit, with the strict consideration of data protection rules. Descriptive statistics will be applied for the variables, and no hypothesis is tested.

National Health Insurance Fund's prescribing and in/outpatient database will be used for the analysis. The database is nationwide, electronic and includes all treated patients. The National Health Insurance Fund provides access to the database to run predefined algorithm. The database is owned by the National Health Insurance Fund.

Descriptive statistics will be applied for the variables. This includes means, median, range, percentage etc. The data of all patients treated with tyrosine kinase inhibitors for chronic myeloid leukemia in Hungary will be studied.

# 9.7. Data analysis

Descriptive statistics will be applied for the variables. This includes means, median, range, percentage etc. The data of all patients treated with tyrosine kinase inhibitors for chronic myeloid leukemia in Hungary will be studied.

Hungary provides universal healthcare for its citizens, thanks to the single-payer public system, the NHIF database contains all prescription claims data of all reimbursed medicinal products, all outpatient and inpatient data from all Hungarian patients.

For the analysis we use electronically stored data from the NHIF database, which display demographic data, previous treatments' and concurrent treatments' data, coded by ICD-10, ICHI and drug TTT codes using a predefined algorithm. Data are provided in anonymized form by the NHIF.

The demographics, treatment lines and treatment sequences with tyrosine kinase inhibitors will be investigated. Patients' comorbidities will also be investigated.

- 1. Epidemiology: age, sex, treatment lines, incidence, prevalence, mortality. For studying the epidemiology based on the NHIF database the following definitions will be used:
  - Patient population is defined as patient is coded with ICD-10 C92 between January 2009 and June 2020, has data either in outpatient or in inpatient system and/or have a TKI (imatinib, bosutinib, dasatinib, nilotinib or ponatinib) prescribed. The analysis period defined as January 2011- June 2020 (January 2009-December 2010 used as pre-exploratory period.)
  - Incidence is defined as patients newly diagnosed during a given period.
  - Point prevalence is defined as patients who were already diagnosed before the first day of the given period (up to 31 December 2008) and were still living on the first day of the given period. They are patients who are still diagnosed on the first day of the given period (cross-sectional view).
  - Period prevalence is defined as patients who were already diagnosed before the
    first day of the given period (up to 31 December 2008) or were newly diagnosed
    during a given period and were still living on the first day of the given period.
    They are the sum of incident and point prevalent patients (longitudinal-section
    view).
  - Dead patient is defined as patient who was diagnosed before the first day of the given period (up to and including 31 December 2008) or during the given period and died during the given period.

- Number of patients treated: patients who were diagnosed and also received TKI treatment at least once during the investigated period, and the TKI treatment was prescribed with C92 ICD-10. The data are also presented in line setting: the first target product (TKI) received is the 1st line treatment, the second target product (TKI) is the 2nd line treatment, and so on.
- 2. Length of each treatment line, overall survival (OS)
  - Medication (TKIs) persistence will be analyzed in the whole investigated population and based on treatment lines. Patients will be enrolled who had first prescription of TKI during the investigated period. Data will be available both censored at death and not censored. Median and 95% CI will also be used to calculate persistence.
    - Persistence of the target product: the patient's therapy is stopped when the target product (TKI) is depleted according to our calculations
    - Persistence of total CML therapy: the patient's therapy is stopped when the patient uses none of the target product (TKI)
  - Length of treatment line will be calculated and demonstrated with Kaplan-Meier curve. Progression considered as change of therapy line or death.
  - Switch in treatment lines determined when the prescribed TKI for CML changed. Therapy switch can be established due to suboptimal treatment response, treatment failure or treatment intolerance. The background of the TKI switch cannot be analyzed using the NHIF's database.
  - Overall survival rate: the probability that a patient is still alive for a certain period of time (% of patients). OS will be demonstrated with Kaplan-Meier curve. The method provides information on the survival of patients in a particular sequence of treatment. Patients will be enrolled who had first prescription of TKI during the investigated period.
    - Overall survival by treatment sequences, as defined in Table 1. based on the actual marketing authorization of the target TKIs

**Table 1. Treatment sequence options.** 

| | 1L | 2L | 3L | 4L | 5L |
|---|----------|-----------|-----------|-----------|-----------|
| 1 | 2 | dosotinih | bosutinib | ponatinib | |
| 2 | | nilatinih | dasatinib | ponatinib | bosutinib |
| 3 | imatinib | nilotinib | | dasatinib | bosutinib |
| 4 | | ponatinib | bosutinib | dasatinib | |

| 5 | | | bosutinib | dasatinib | ponatinib |
|----|---------------------|------------|-----------|-----------|-----------|
| 6 | | | | ponatinib | dasatinib |
| 7 | 8<br>9<br>dasatinib | docatinih | nilotinib | bosutinib | ponatinib |
| 8 | | | | ponatinib | bosutinib |
| 9 | | | bosutinib | nilotinib | ponatinib |
| 10 | | uasatiiiib | | ponatinib | nilotinib |
| 11 | | ponatinib | bosutinib | nilotinib | |
| 12 | | | nilotinib | bosutinib | |
| 13 | | bosutinib | nilotinib | dasatinib | ponatinib |
| 14 | | | | ponatinib | dasatinib |
| 15 | | | dasatinib | ponatinib | dasatinib |
| 16 | | | | nilotinib | ponatinib |
| 17 | | dasatinib | bosutinib | ponatinib | |
| 18 | | uasatiiiib | ponatinib | bosutinib | |
| 19 | | bosutinib | dasatinib | ponatinib | |
| 20 | 1 dasatinib | nilotinib | bosutinib | ponatinib | |
| 21 | | | ponatinib | bosutinib | |
| 22 | | bosutinib | nilotinib | ponatinib | |
| 23 | 23 other | | | | |

Table 1. contains predefined treatment sequence options based on the products EMA label. However real-world sequences may differ due to the reimbursement, NPP, etc. in Hungary. Other defined as all other sequence not listed in the table and will be detailed based on the results of the analysis.

- 3. Comorbidities (based on Charlson comorbidity index<sup>10</sup>), number of comorbidities on each line:
  - We determine what comorbidities existed in patients at the time of diagnosis of CML. In addition, the distribution of CML patients without comorbidity, with 1 or 2 or more comorbidities will be analyzed.
  - Investigation of the comorbidities is based on the Charlson comorbidity index as following:

## **Table 2. Definitions of comorbidities**

| Condition | Definition upon ICD-10 |
|---|---|
| Ischemic heart disease | I2000-I2590 |
| Congestive heart failure | I50 |
| Arrythmiac condition (including AF) | I44, I45, I47, I48, I49 |
| Hypertonia | I10, I11, I12, I13, I15 |
| Peripheral vascular disease | I70, I73, R02, Z958, Z959 |
| Cerebral vascular accident | I60, I61, I62, I63, I65, I66, G450, G451, G452, G458, G459, G46, I64, G454, I670, I671, I672, I674, I675, I676, I677 I678, I679, I681, I682, I688, I69 |
| Dementia | F01, F02, F03, F051 |
| Pulmonary disease (lower tract) | J4 |
| Connective tissue disorder | M32, M34, M332, M053, M058, M059, M060, M063, M069, M050, M052, M051, M353 |
| Peptic ulcer | K25, K26, K27, K28 |
| Liver disease | K7 |
| Severe liver disease | K729, K766, K767, K721 |
| Diabetes | E10-14 |
| Diabetes complications | E102, E112, E132, E142 E103, E113, E133, E143 E104, E114, E134, E144 |
| Paraplegia | G81 G041, G820, G821, G822 |
| Renal disease | N03, N052, N053, N054, N055, N056, N072, N073, N074, N01, N18, N19, N25 |
| Other cancer | С |
| Metastatic cancer | C77, C78, C79, C80 |
| HIV | B20, B21, B22, B23, B24 |
| Thromboembolic events | I26, I800-I8290 |
| Metabolic disorders | E7800, E7810, E7820, E7830, E7840, E7850, E10-E14, |

4. Dose intensity: The average doses of the investigated TKIs will be analysed by therapeutic lines regardless of the previous and following treatment.

# 9.8. Limitations of the research methods

Since the NHIF database only contains reimbursed prescription claims data, non-reimbursed claims (e.g. clinical trial patients or privately reimbursed treatment which is uncommon in

Hungary). The database does not contain laboratory data (e.g. neutropenia, anemia, etc.), patient parameters (e.g. body mass index), patient symptoms (e.g. fatigue) or pathological or molecular features of CML (depth of treatment response g. CCR, MR, MR4.0, MR4.5, etc.) The database does not contain information on adverse events. The database does not include data on the background of therapy switch (suboptimal treatment response, treatment failure or treatment intolerance) hence the progression free interval cannot be investigated only the length of therapy per lines.

#### **Biases:**

Selection bias: Given the retrospective data collection, the study population enrolled in this study is based on treating physician clinical decision and selection.

*Information bias:* Data provided by the NHIF database based on electronic health records coded, thus it has limitations, and certain information of pathological or molecular features of CML is not coded.

## 9.9. Other aspects

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 10.2. Patient consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

# 10.3. Institutional review board (IRB)/Independent ethics committee (IEC)

There must be prospective approval of the study protocol, protocol amendments, and other relevant documents (e.g., informed consent forms if applicable) from the relevant IRBs/IECs. All correspondence with the IRB/IEC must be retained. Copies of IRB/IEC approvals must be forwarded to Pfizer.

The study protocol approved by Hungarian National Institute of Pharmacy and Nutrition, and by Medical Research Council Ethical Committee

# 10.4. Ethical conduct of the study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor.

The study protocol approved by Hungarian National Institute of Pharmacy and Nutrition, and by Medical Research Council Ethical Committee.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start.

In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

Hungarian DSU is informed about the study.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable competent authority in any area of the world, or if the party responsible for collecting data from the participant (RxTarget Statistical Programming and Analysis Ltd.) is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

Peer reviewed journal publication is planned with the authorship of the investigators and statistics partner.

#### 13. REFERENCES

- 1. Demeter J. et al. A krónikus myeloid leukémia korszerű diagnosztikája és kezelése Orvosi Hetilap Volume 157: Issue 37 https://doi.org/10.1556/650.2016.30521
- 2. Hochhaus A et al. European LeukemiaNet 2020 recommendations for treating chronic myeloid leukemia Leukemia 2020 https://doi.org/10.1038/s41375-020-0776-2
- 3. Gaál-Weisinger et al. Újdonságok és tapasztalatok a krónikus mieloid leukémia tirozinkináz-gátló kezelésében; Magyar Onkológia 61:67–74, 2017
- 4. Pfirrmann et al. Prognosis of long-term survival considering disease-specific death in patients with chronic myeloid leukemia; Leukemia volume 30, pages48–56(2016)
- 5. García-Gutiérrez et al. Tyrosine Kinase Inhibitors Available for Chronic Myeloid Leukemia: Efficacy and Safety Front Oncol. 2019; 9: 603
- 6. Breccia et al. How many chronic myeloid leukemia patients who started a frontline second-generation tyrosine kinase inhibitor have to switch to a second-line treatment? A retrospective analysis from the monitoring registries of the italian medicines agency (AIFA); Cancer Medicine. 2020;00:1–6.

- 7. Hoffman et al, The EUTOS population-based registry: incidence and clinical characteristics of 2904 CML patients in 20 European Countries; Leukemia (2015) 29, 1336–1343
- 8. 31/2010. (V. 13.) EüM rendelet a finanszírozási eljárásrendekről 2020. https://net.jogtar.hu/getpdf?docid=A1000031.EUM&targetdate=fffffff4&printTitle= 31/2010.+%28V.+13.%29+E%C3%BCM+rendelet&referer=http%3A//net.jogtar.hu/jr/gen/hjegy doc.cgi%3Ffdocid%3D00000001.TXT
- 9. García-Gutiérrez et al. Tyrosine Kinase Inhibitors Available for Chronic Myeloid Leukemia: Efficacy and Safety Front Oncol. 2019; 9: 603.
- 10. Sundararajan et al. New ICD-10 version of the Charlson Comorbidity Index predicted in-hospital mortality Journal of Clinical Epidemiology 57 (2004) 1288–1294

## 14. LIST OF TABLES

Table 1. Treatment sequence options.

Table 2. Definitions of comorbidities

## 15. LIST OF FIGURES

Figure 1. Study design

ANNEX 1. LIST OF STAND ALONE DOCUMENTS

None

**ANNEX 2. ADDITIONAL INFORMATION** 

Not applicable.